CLINICAL TRIAL: NCT07145736
Title: Moxidectin Versus Ivermectin as Mass Drug Administration for the Control of Onchocerciasis and Other Neglected Tropical Diseases: A Cluster-randomised Trial
Brief Title: Moxidectin Versus Ivermectin as Mass Drug Administration for the Control of Onchocerciasis and Other Neglected Tropical Diseases
Acronym: EKAIO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Emory University (Other); La Trobe University (Other); Murdoch Childrens Research Institute (Other); Medicines Development for Global Health (Other); University of Melbourne (Other); Swiss Tropical & Public Health Institute (Other); University of Ottawa (Other); The Mentor Initiative (Other); Erasmus Medical Center (Other); Ministry of Health, Angola (Unknown); The END Fund (Unknown); Center for Research on Filariasis and Other Tropical Diseases, Cameroon (Other); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KirbyI
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Onchocerciasis; Ascaris Lumbricoides Infection; Trichuris Trichiura; Infection; Hookworm Infections; Scabies
MeSH Terms: conditions — Onchocerciasis; Trichuriasis; Hookworm Infections; Scabies | interventions — moxidectin; Ivermectin

STUDY DESIGN:
Intervention Model Description: Clusters of villages are assigned to either ivermectin or moxidectin in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Moxidectin (Experimental): Single oral dose of moxidectin treatment 8 mg (4 tablets of 2 mg of moxidectin), once per year
  Interventions: Drug: Moxidectin
- Ivermectin (Active Comparator): Single oral dose of ivermectin treatment with approximately 150 µg/kg determined based on height (between 1 and 4 tablets of 3 mg of ivermectin), once per year
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Moxidectin — 2 mg tablets
  Arms: Moxidectin
Drug: Ivermectin — 3 mg tablets
  Arms: Ivermectin

SUMMARY:
This clinical trial compares two treatments - ivermectin and moxidectin - to learn which is better at reducing the proportion of people with onchocerciasis (river blindness) when given through mass drug administration (MDA) in Angola. Both drugs are approved by the United States Food and Drug Administration (FDA) to treat this disease. The study also explores how these treatments affect other infections common in the region, including intestinal worms (soil-transmitted helminths) and scabies.

The trial aims to answer the following key questions:

* How do moxidectin and ivermectin compare in reducing the prevalence (how common the disease is) and intensity (amount of parasites per person) of onchocerciasis in the community?
* Do the treatments differ in their effect on the prevalence and intensity of soil-transmitted helminths and the prevalence of scabies?
* Does moxidectin reduce transmission of onchocerciasis more effectively than ivermectin, based on genetic testing of parasites in people and lab testing of the blackflies that carry the infection?
* How many more years of treatment would be needed to reach elimination with each drug, based on mathematical disease modelling?
* How do communities feel about receiving moxidectin versus ivermectin, and what factors help or make it harder to carry out MDA programs with moxidectin versus ivermectin?

The study takes place in Bié Province, Angola, and involves 20 groups of villages randomly assigned to receive either moxidectin or ivermectin once a year for four years. Prior to every round of MDA, researchers will collect skin, stool and blood samples from a sample of the people living in the study area. We believe the results will help guide global policy on the use of moxidectin in efforts to eliminate onchocerciasis and control related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children and adults
* Residents in the villages selected for MDA treatment

Exclusion Criteria:

* Arm 1 (ivermectin): children under the age of 5 and/or under 90 cm of height
* Arm 2 (moxidectin): children under the age of 12 years (who will receive ivermectin if they are at least 90 cm in height/5 years of age and above).
* Arm 1 (ivermectin): Women breast-feeding babies under 45 days of age
* Arm 2 (moxidectin): All breastfeeding women (who will be offered ivermectin if their infants is at least 45 days old)
* Know allergy to ivermectin or moxidectin
* Attending other clinical trials during the study
* Pregnant
* Arm 2 (moxidectin): Women planning to become pregnant in the 3 months post-treatment
* Refusal to receive one or both study drugs, i.e. participants in villages allocated to receive moxidectin who refuse to receive moxidectin will be given the option to receive ivermectin; if they refuse to receive both drugs they will be excluded from the MDA altogether
* Has an illness that makes them too sick or weak to get out of bed
* Currently hospitalized

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52000 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Onchocerca volvulus microfilariae | 36 months after the first intervention
  Prevalence of O. volvulus microfilariae at 36 months in skin snips, the marker most likely to show change in the shorter term as demonstrated by the therapeutic trials

SECONDARY OUTCOMES:
Prevalence of O. volvulus microfilaria/mg skin | 12, 24 and 36 months after the first intervention
Microfilariae density (mean, median) | 12, 24 and 36 months after the first intervention
Prevalence of nodules | 12, 24 and 36 months after the first intervention
Prevalence of onchocerciasis skin disease | 12, 24 and 36 months after the first intervention
Proportion of black flies with infective O. volvulus larvae | 12, 24 and 36 months after the first intervention
  Infection assessed based on all 3 are markers recommended by WHO to define population-level elimination
Prevalence of anti-Ov-16 | 12, 24 and 36 months after the first intervention
Prevalence of Ascaris lumbricoides | 12, 24 and 36 months after the first intervention
  Measured through qPCR
Intensity of Ascaris lumbricoides infection | 12, 24 and 36 months after the first intervention
  Measured through qPCR
Prevalence of Trichuris trichiura | 12, 24 and 36 months after the first intervention
  Measured through qPCR
Intensity of Trichuris trichiura infection | Baseline and 12, 24 and 36 months after the first intervention
  Measured through qPCR
Prevalence of hookworm | 12, 24 and 36 months after the first intervention
  Measured through qPCR
Intensity of hookworm infection | 12, 24 and 36 months after the first intervention
  Measured through qPCR
Prevalence of Strongyloides stercoralis | 12, 24 and 36 months after the first intervention
  Measured through qPCR
Intensity of Strongyloides stercoralis infection | 12, 24 and 36 months after the first intervention
  Measured through qPCR
Prevalence of scabies/impetigo | 12, 24 and 36 months after the first intervention

CONTACTS AND LOCATIONS:
Overall Officials: Susana V Nery, PhD, Principal Investigator — Kirby Institute, University of New South Wales, Australia
Locations (1):
- Villages in Andulo and Nharea Municipalities, Andulo, Bíe Province, Angola

IPD SHARING:
Plan to Share IPD: Undecided